CLINICAL TRIAL: NCT06056102
Title: Autologous Chimeric Antigen Receptor Engineered T Cell Immunotherapy for Desensitization in Patients Awaiting Kidney Transplantation
Brief Title: CAR-T Cell Therapy for Desensitization in Kidney Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Pennsylvania Clinical Cell and Vaccine Production Facility (CVPF) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-46
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant; Kidney Failure; End Stage Renal Failure on Dialysis
Keywords: Kidney transplant; CART-BCMA; huCART-19; Highly sensitized; cPRA; UNOS waiting list; End stage renal failure patients with cPRA >99.5%
MeSH Terms: conditions — Renal Insufficiency | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participant Cohorts (Experimental): * Safety Run-in phase (2 subjects at UPenn)
  * Cohort 1 (3-6 subjects)
  * Cohort 2 (3-6 subjects)
  * Cohort 3 (3-6 subjects)
  Interventions: Drug: Cyclophosphamide; Biological: CART-BCMA; Biological: huCART19; Drug: Fludarabine

INTERVENTIONS:
Drug: Cyclophosphamide — * Safety Run-in: 375mg/m^2 daily x 3
  * Cohort 1: 375mg/m^2 daily x 3
  * Cohort 2: 375mg/m^2 daily x 3
  * Cohort 3: 375mg/m^2 daily x 3
  Other Names: Cytoxan
Biological: CART-BCMA — * Safety Run-in: 5 x 10^7 CAR T cells
  * Cohort 1: 1.5 x 10^8 CAR T cells
  * Cohort 2: 1.5 x 10^8 CAR T cells
  * Cohort 3: 5 x 10^8 CAR T cells
  Other Names: Chimeric Antigen Receptor T cell (CART)/B cell maturation antigen (BCMA)
Biological: huCART19 — * Safety Run-in: 5 x 10^7 CAR T cells
  * Cohort 1: 1.5 x 10^8 CAR T cells
  * Cohort 2: 1.5 x 10^8 CAR T cells
  * Cohort 3: 5 x 10^8 CAR T cells
  Other Names: Chimeric Antigen Receptor T cell (CART)/ CD-19 Targeted Humanized CAR T Cell
Drug: Fludarabine — • Cohort 3: 24mg/m^2 daily x 3
  Other Names: Fludara

SUMMARY:
This research study is for people who have been waiting for a kidney transplant for at least one year, and who have a cPRA of 99.5% or higher. Having a cPRA of 99.5% or higher means that your immune system would reject 99.5% of kidneys available for transplant. The study will test whether new products called Chimeric Antigen Receptor T Cells (CAR T Cells), when given with chemotherapy, is safe and will reduce cPRA.

The main study will last up to 2 years: Participants will have up to 30 clinic or hospital visits over a one-year period. If a transplant takes place, there will be 9 more visits after transplant. Long term follow up is required by the Food and Drug Administration (FDA) for 15 years after receiving CAR T cell.

The primary objective is to evaluate the safety and feasibility of administering CART BCMA + huCART-19 following lymphodepletion, including determination of optimal tolerated regimen (OTR) and/or recommended phase 2 regimen, according to the incidence of dose limiting toxicity (DLT) in highly sensitized patients awaiting kidney transplant.

DETAILED DESCRIPTION:
CTOT-46 will enroll up to up to 20 highly sensitized kidney transplant candidates at 3 centers. There will be a safety run-in and 3 treatment cohorts to assess the safety and pharmacodynamics of CART-BCMA and huCART-19.

Following screening and enrollment, the subject will undergo leukapheresis to collect T cells for CAR T cell manufacturing. Subsequently, subjects will undergo lymphodepleting chemotherapy followed by CART-BCMA and huCART19 cell infusions. A secondary objective is to evaluate the efficacy of study treatment to reduce cPRA and determine the duration cPRA reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-65 years with kidney failure requiring hemodialysis.
2. United Network for Organ Sharing (UNOS) listed for kidney transplant for at least 1 year.
3. Patients must meet one of the following two criteria:

   1. Protocol-specific cPRA ≥99.5-99.895% AND no matched living donor, ineligible for kidney paired donation programs, have blood group Type O or B, have documentation of virtual crossmatch (current or past) and predictive of a positive physical crossmatch to a deceased donor
   2. Protocol-specific cPRA ≥99.9% Protocol-specific cPRA must be rounded from three significant figures measured ≤90 days from the time of enrollment (i.e., cPRA of 0.994500 or 0.998500 would be eligible) using the web-based OPTN cPRA calculator (https://optn.transplant.hrsa.gov/resources/allocation-calculators/cpra-calculator/); accounting for HLA-A, -B, -C, -DRB1, -DRB3/4/5, and -DQB1 Luminex Single Antigen Beads (SAB) with MFI ≥3000; 1 archived sample within 6 months of screening required.
4. Based on center-specific listing policies, a cPRA in UNet Waitlist that is ≥99.5% (the candidate must be eligible for additional priority of kidneys equivalent to individuals with a 100% cPRA)
5. Able to understand and give written informed consent to participate in all aspects of the study.
6. Willing to stay within 2 hours of the home study site for at least 28 days after the last T cell infusion
7. Subjects of reproductive potential must agree to use contraception for at least one year after CAR T Cell infusion
8. In the absence of contraindication, vaccinations must be up to date per the DAIT Guidance for Patients in Transplant Trials and include TdAP
9. Positive for EBV capsid IgG
10. Negative testing for latent TB infection within 3 months prior to enrollment. Testing should be conducted using either a PPD or interferon-gamma release assay (i.e. QuantiFERON-TB, T-SPOT.TB). Patients with a positive test for latent TB infection must complete appropriate therapy for Latent Tuberculosis Infection (LTBI). A subject is considered eligible only if they have a negative test for LTBI within 3 months prior to enrollment OR they have appropriately completed LTBI therapy prior to transplant. Latent TB infection treatment regimens should be among those endorsed by the CDC
11. Hemoglobin ≥9g/dL
12. ANC ≥ 1,800/μL, > 1,200/ μL for patients with Duffy-null associated neutrophil count (DANC)
13. Absolute Lymphocyte Counts ≥500/μL or CD3 T cell Count ≥150/μL
14. Platelet count ≥120,000/μL

Exclusion Criteria:

1. Subjects with indwelling catheters as primary access for hemodialysis
2. Previous solid organ (except kidney) or bone marrow transplant
3. BMI ≥35 kg/m^2
4. Subjects who have preserved or oliguric urine output > 100 cc/day with history of recurrent UTI (2 in 6 months or 3 in 1 year, see study definitions)
5. Subjects described in exclusion #4 with structural disease such as polycystic kidney disease, obstructive uropathy with nephrolithiasis or those otherwise at higher risk of urinary tract infections. Anuric subjects with structural kidney disease are not excluded
6. Known active current or history of invasive fungal infection; any non-tuberculous mycobacterial infection that has been active or has required therapy within the last year. Any infection requiring hospitalization and IV antibiotics within 4 weeks of screening or PO antibiotics within 2 weeks
7. History of HIV, chronic HBV, or chronic HCV, regardless of treatment
8. Negative CMV serology
9. Detectible viral load HBV, HCV, CMV, EBV, or BK by PCR
10. Any B cell depleting or monoclonal antibody therapy within 6 months prior to enrollment
11. Receiving ongoing immunosuppression including corticosteroids, intravenous immunoglobulin, cyclophosphamide, tacrolimus, mycophenolic acid, or azathioprine from 90 days prior to study entry
12. Active auto-immune disease, including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis, or have a history of severe (as judged by the investigator) autoimmune disease requiring prolonged immunosuppressive therapy, except for renal-limited autoimmune conditions without risk for systemic manifestations (e.g. IgA nephropathy)
13. Any chronic illness requiring uninterrupted anti-coagulation or anti-platelet therapy
14. History of cirrhosis or severe liver disease, including abnormal liver profile (aspartate aminotransferase [AST], alanine aminotransferases [ALT] or total bilirubin > 3 times upper limit of normal at screening (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome)
15. History of sickle cell disease, or systemic amyloidosis
16. Cardiac clearance for transplant > 6 months old and/or any of the following: NYHA Class III or IV heart failure, unstable angina, left ventricular ejection fraction < 40%, a history of recent (within 6 months) myocardial infarction or implantable cardioverter/ defibrillators and/or biventricular pacing.
17. Moderate-severe pulmonary function abnormality, defined as resting oxygen saturation <92% on room air or FEV1, TLC, or DLCO (after correction for hemoglobin) <50% of predicted values
18. Patients who have received any live vaccine within 30 days of planned leukapheresis
19. Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational drug, whichever is longer) of screening
20. Pregnant, currently breastfeeding, or planning to become pregnant during the primary or post-transplant follow up of the study.
21. Past or current social or medical problems; or findings from physical examination or laboratory testing that are not listed above, which in the opinion of investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Lymphodepleting Chemotherapy Eligibility:

Study entry eligibility must be re-assessed prior to starting lymphodepletion. In addition, subjects must undergo respiratory viral testing on nasal or nasopharyngeal swabs (per institutional practice) for SARS-CoV-2 and influenza within 7 days prior to the first planned lymphodepletion chemotherapy.

1. If the subject is positive for influenza, Tamiflu® or equivalent should be administered per package insert. The subject must complete treatment and symptoms must be improving and either resolved or nearly resolved in the judgment of the treating investigator prior to receiving lymphodepleting chemotherapy and CAR T cells. Repeat influenza testing is not required prior to initiating lymphodepleting chemotherapy and CAR T cell infusion.
2. If the subject tests positive for SARS-CoV-2, the subject will be managed per institutional practice. Subject will be eligible to initiate lymphodepleting chemotherapy and CAR T cell infusion once cleared from requirement for isolation according to institutional and/or CDC guidance.
3. If testing is positive for another respiratory virus (e.g., as part of a multiplex respiratory pathogen panel in the course of testing for influenza or SARS-CoV-2), the lymphodepleting chemotherapy and CAR T cell infusion will be delayed for at least 7 days to be sure clinical symptoms of a viral infection do not develop. If clinical symptoms develop, the lymphodepleting chemotherapy and CAR T cell infusion will be delayed until resolution of these symptoms.

CAR T Cell Infusion Eligibility:

The criteria below will be assessed by the investigator following lymphodepleting chemotherapy and before administration of CAR T cells. Subjects who do not satisfy these criteria may have CAR T cell infusion delayed until such time as criteria are satisfied. Subjects who receive lymphodepleting chemotherapy but in whom CAR T cell infusion is delayed >4 weeks after the first day of lymphodepleting chemotherapy will receive a second cycle of lymphodepleting chemotherapy prior to CAR T cell infusion. For subjects receiving fludarabine, a second cycle of cyclophosphamide can be administered, but fludarabine will not be repeated.

1. Subjects must not have developed deterioration in performance status or overall clinical condition or new laboratory abnormalities that would, in the opinion of the treating investigator, render it unsafe to proceed with CAR T cell infusion. The following are specific conditions that warrant delaying CAR T cell infusion:

   1. Requirement for supplemental oxygen to maintain peripheral oxygen saturation ≥95%.
   2. Presence of clinically significant radiographic abnormalities on chest x-ray. Chest x-ray is not required to evaluate for radiographic abnormalities in the absence of suggestive symptoms or exam findings.
   3. New cardiac arrhythmia not controlled with medical management. EKG is not required to evaluate for arrhythmia in the absence of suggestive symptoms or exam findings.
   4. Hypotension requiring vasopressor support.
   5. Active infection: Diagnostic test results indicating new bacterial, fungal, or viral infection within prior 48 hours.
2. Subjects must have adhered to restrictions on pre-infusion therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2042-12-15 (Estimated)

PRIMARY OUTCOMES:
The timing of adverse events after infusion of Chimeric antigen receptor T - B cell maturation antigen (CART-BCMA) with CD19 Targeted Humanized CAR T Cell (huCART-19) | From time of lymphodepletion to 12 months
  Adverse events will be categorized and described according to CTCAE v5.0. Specific safety outcomes will include but are not limited to:
  1. Cytokine release syndrome, as defined by American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
  2. Neurotoxicity (ICANS), as defined by ASTCT consensus grading
  3. Delayed hematopoetic recovery: proportion of subjects achieving ANC >1,000/microL and Platelets >75,000/microL at 60 days after first CART cell infusion
  4. Dose limiting toxicity
The frequency of adverse events after infusion of Chimeric antigen receptor T - B cell maturation antigen (CART-BCMA) with CD19 Targeted Humanized CAR T Cell (huCART-19) | From time of lymphodepletion to 12 months
  Adverse events will be categorized and described according to CTCAE v5.0. Specific safety outcomes will include but are not limited to:
  1. Cytokine release syndrome, as defined by ASTCT consensus grading
  2. Neurotoxicity (ICANS), as defined by ASTCT consensus grading
  3. Delayed hematopoetic recovery: proportion of subjects achieving ANC >1,000/microL and Platelets >75,000/microL at 60 days after first CART cell infusion
  4. Dose limiting toxicity
The severity of adverse events after infusion of Chimeric antigen receptor T - B cell maturation antigen (CART-BCMA) with CD19 Targeted Humanized CAR T Cell (huCART-19) | From time of lymphodepletion to 12 months
  Adverse events will be categorized and described according to CTCAE v5.0. Specific safety outcomes will include but are not limited to:
  1. Cytokine release syndrome, as defined by ASTCT consensus grading
  2. Neurotoxicity (ICANS), as defined by ASTCT consensus grading
  3. Delayed hematopoetic recovery: proportion of subjects achieving ANC >1,000/microL and Platelets >75,000/microL at 60 days after first CART cell infusion
  4. Dose limiting toxicity
The proportion of apheresed subjects who receive the intended/planned Chimeric antigen receptor T (CAR T) cell dose in the respective cohort | From time of lymphodepletion to 12 months

SECONDARY OUTCOMES:
The proportion of subjects meeting the predefined Calculated Panel Reactive Antibody (cPRA) reduction criteria after the infusion of CART-BCMA + huCART-19 | 26 weeks after the infusion
Duration of Calculated Panel Reactive Antibody (cPRA) response | From time of infusion to 12 months
For subjects who are transplanted, the proportion of subjects experiencing acute cellular rejection or antibody mediated rejection, delayed graft function (as well as AKI), graft loss OR De Novo donor specific antibody | 3 years after transplantation
The proportion of subjects with opportunistic infections | From time of infusion to 12 months or 3 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Bhoj, M.D., Ph.D., Study Chair — University of Pennsylvania Medical Center: Transplantation; Ali Naji, MD, Ph.D., Principal Investigator — University of Pennsylvania Medical Center: Transplantation; Alfred Garfall, MD, Study Chair — University of Pennsylvania Medical Center: Transplantation
Locations (3):
- United States (3):
  - Massachusetts General Hospital: Transplantation (Site #: 71107), Boston, Massachusetts
  - NYU Langone Health (Site #: 71177), New York, New York
  - University of Pennsylvania Medical Center (Site #: 71111), Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Vo A, Ammerman N, Jordan SC. New Therapies for Highly Sensitized Patients on the Waiting List. Kidney360. 2024 Aug 1;5(8):1207-1225. doi: 10.34067/KID.0000000000000509. Epub 2024 Jul 12. PMID 38995690